CLINICAL TRIAL: NCT04988334
Title: Improving Capacity to Reduce Fall-Related Injury Risk in Older Adults
Acronym: FAST2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other); Saskatchewan Centre for Patient-Oriented Research (Other)
Responsible Party: Principal Investigator, Cathy Arnold, Professor, University of Saskatchewan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: University of Saskatchewan
Record Dates: First submitted 2021-07-28; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Fall Injury

STUDY DESIGN:
Intervention Model Description: wait list control to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAST (Active Comparator): 12 weeks of FAST, 2/week 45 minute sessions with half hour per week of education, same group of men and women
  Interventions: Other: Wait Control
- wait control (Placebo Comparator): 12 weeks of usual activity prior to intervention, same group of men and women
  Interventions: Other: Wait Control

INTERVENTIONS:
Other: Wait Control — usual activities

SUMMARY:
Fall Arrest Strategy Training (FAST) is a unique, simple exercise program designed to improve one's ability to prevent injury when a fall is unavoidable. Women are more likely to participate in fall prevention programming than men despite risk of serious fall related injuries such as head injury similar in both men and women. The purpose of this project is to test differences between men and women's physical capacity to control the downward descent of a forward fall and prevent injury and to understand factors that influence participation of women and men in fall prevention programming. A total of 60 seniors (30 men and 30 women) age 60 years or older will do their regular activities for 12 weeks followed by 12 weeks of FAST training. They will be tested before and after for muscle strength, balance and their ability to land and descend in a simulated forward fall using a safe protocol in our lab. Group discussions among women and men after FAST will help us determine facilitators and barriers to exercise participation.

DETAILED DESCRIPTION:
The purpose of this proposed study is to advance our knowledge of this innovative and simple training program, FAST, to determine if it has potential to improve the physical capacity to arrest a fall and reduce injury risk in older community-dwelling women and men. Using our novel lab-based energy absorption and strength measures, we will be able to compare fall-arrest capacity changes in older men and women.This study will also help to inform strategies to engage older men in exercise programming.

Research Goals and Objectives: The principal research questions of this study are:

1. Does the FAST improve fall arrest capacity in older women and men as compared to usual activity (wait control period)?,
2. Does FAST increase arm muscle strength, response time, mobility and balance control compared to usual activity? ,
3. Are there sex differences in fall risk changes, fall arrest capacity, and chance of head impact? and
4. Do men differ from women in their perceptions of the barriers and facilitators to participating in FAST? The hypotheses are that: 1) FAST will result in greater improvements in energy absorption, UE strength, response time and mobility compared to usual activity for both older men and women; however 2) men will demonstrate enhanced fall arrest capacity and 3) will identify unique barriers and facilitators to participation compared to women.

The study is a quasi-experimental pre-post design with a wait list control period where 60 men and women, age 60 years or older will be recruited to participate in FAST.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years living in the community

Exclusion Criteria:

* recent upper body injury or pain,
* recent or history of more than one distal radial fracture,
* history of upper extremity neurological conditions or conditions contradicting upper extremity strength testing or training,
* signs of severe cognitive impairment identified with the mini-Cog
* unable to safely ambulate independently in the community

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Muscle strength dynamic | 12 weeks
  concentric and eccentric isokinetic dynamometry
Muscle Strength isometric | 12 weeks
  Hand held dynamometry
Muscle Strength isometric | 12 weeks
  grip strength
Muscle strength isometric | 12 weeks
  push off test
response time | 12 weeks
  signal to touch on force plate
Balance | 12 weeks
  one leg stand
Balance | 12 weeks
  tandem stand
Balance | 12 weeks
  modified clinical test of sensory interaction and balancer
Balance Confidence | 12 weeks
  Activities balance confidence scale
Fall Risk | 12 weeks
  Fall Risk for older people in the community-screen
timed up and go test | 12 weeks
  stand, walk 3 meters, turn and return to sit
chair stand | 12 weeks
  30-second chair stand test
gait velocity | 12 weeks
  timed 6 meters within 10 meter walk
fall landing capacity | 12 weeks
  energy absorption, force, elbow range of motion

OTHER OUTCOMES:
physical activity | 12 weeks
  physical activity scale for the elderly
fall history | 12 weeks
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Cathy o Arnold, Principal Investigator — School of Physical Therapy
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Undecided
de-identified group data to be shared via peer review publication and on request to corresponding author